CLINICAL TRIAL: NCT07326605
Title: Discriminative and Prognostic Value of Myocardial Energetics and Pressure-Volume Loop Parameters Derived From Cardiac MRI in Heart Failure With Preserved Ejection Fraction
Brief Title: Cardiac MRI-Derived Pressure-Volume Loop Analysis in Heart Failure With Preserved Ejection Fraction
Acronym: CMR-PV HFpEF
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, MD, PhD, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CMR-PV HFpEF; 82471973 (Other Grant/Funding Number: National Natural Science Foundation of China); 7242110 (Other Grant/Funding Number: Beijing Natural Science Foundation); 3332025134 (Other Grant/Funding Number: Fundamental Research Funds for the Central Universities)
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: Cardiac MRI; Heart failure with preserved ejection fraction; Pressure loop analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFpEF patients: Heart failure with preserved ejection fraction (HFpEF) patients
- Healthy controls: Sex- and age-matched healthy controls

SUMMARY:
This is a multi-center, observational study designed to evaluate the discriminative and prognostic value of pressure-volume (PV) loop analysis parameters and myocardial energetics derived from cardiac MRI in patients with heart failure with preserved ejection fraction (HFpEF). This study plans to enroll 3000 adult HFpEF patients and 500 adult healthy controls. The primary clinical endpoint was a composite of all-cause mortality and heart failure hospitalization, with events ascertained through medical records, clinic visits, and telephone follow-up. This study aims to determine whether cardiac MRI-derived PV loop analysis parameters and myocardial energetics provide incremental discriminative and prognostic information beyond conventional cardiac MRI parameters in patients with HFpEF. The study is non-interventional and does not involve any investigational drugs or devices.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms and/or signs of HF ≥ New York Heart Association (NYHA) class II;
2. Left ventricular ejection fraction (LVEF) of 50% or higher;
3. N-terminal fragment of the prohormone of brain natriuretic peptide (NT-proBNP) level > 125 pg/mL or brain natriuretic peptide (BNP) level > 35 pg/mL in sinus rhythm, or NT-proBNP level > 365 pg/mL or BNP level > 105 pg/mL in atrial fibrillation;
4. At least one of objective indicators of (i) cardiac structural abnormalities including LA maximum volume index (LAVi max) > 29 mL/m2 or echocardiography-measured LV end-diastolic mass index (LVMi) ≥ 115 g/m2 for men and ≥ 95 g/m2 for women, and (ii) LV diastolic dysfunction including early and/or late diastolic mitral inflow velocity (E/A) < 1 or early diastolic mitral inflow velocity and/or mitral annular peak early diastolic velocity (E/e') > 13.

Exclusion Criteria:

1. Primary cardiomyopathy;
2. Acute coronary syndrome;
3. Primary severe valvular heart disease;
4. Acute pulmonary embolism;
5. Severe renal dysfunction;
6. Poor image quality that was insufficient to identify myocardial endocardium and epicardium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with preserved ejection fraction experienced cardiac MRI scanning
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with All-Cause Death | 3-year
  All-cause death was defined as death from any cause occurring during the 3-year follow-up period. Mortality status was ascertained through review of medical records, hospital discharge summaries, and follow-up contacts.

SECONDARY OUTCOMES:
Number of Participants with Cardiovascular Death | 3-year
  Cardiovascular death was defined as death resulting from cardiovascular causes occurring during the 3-year follow-up period. Cardiovascular causes included, but were not limited to, myocardial infarction, heart failure, fatal arrhythmia, stroke, or sudden cardiac death. The outcome was ascertained through review of medical records, hospital discharge summaries, and follow-up contacts.
Number of Participants with Heart Failure Hospitalization | 3-year
  Heart failure hospitalization was defined as any hospitalization for heart failure occurring during the 3-year follow-up period. Hospitalizations were identified based on hospital admission records with a primary diagnosis of heart failure.